CLINICAL TRIAL: NCT05755711
Title: Equity in Modifying Plaque Of WomEn With UndeRtreated Calcified Coronary Artery Disease
Acronym: EMPOWER CAD
Status: Active, not recruiting | Type: Observational
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 67712
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Intravascular Lithotripsy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Female subjects referred for percutaneous coronary intervention: Female subjects referred for percutaneous coronary intervention (PCI) with coronary IVL and stenting per standard of care.
  Interventions: Device: Shockwave Medical Coronary IVL System

INTERVENTIONS:
Device: Shockwave Medical Coronary IVL System — Coronary Intravascular Lithotripsy (IVL)

SUMMARY:
Post-market, prospective, multi-center, single-arm observational study to generate real-world clinical evidence associated with coronary IVL in a population of female subjects with calcified coronary artery disease.

DETAILED DESCRIPTION:
Subject population: up to 400 female subjects referred for percutaneous coronary intervention (PCI) with coronary IVL and stenting per standard of care at up to 50 global sites in the US, UK and Europe. Subjects will have clinical follow-up prior to discharge from the index intervention and at 30 days, 1, 2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a non-pregnant female ≥18 years of age
2. The subject meets indications for PCI and stent
3. The subject is scheduled to undergo PCI with coronary IVL and stenting per standard of care for non-stented lesion
4. The subject is willing to comply with protocol-specified follow-up evaluations
5. The subject, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

1. Subjects with known mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation, or is associated with a life expectancy of less than one year
2. Subjects presenting with cardiogenic shock at the time of the index procedure
3. Serious angiographic complication in the target vessel prior to treatment with coronary IVL including-severe dissection (Type D to F), perforation, abrupt closure, persistent slow-flow or persistent no reflow
4. Subject unable to tolerate anticoagulation/antiplatelet therapy per guidelines
5. Subject is enrolled in any study of an investigational device or drug that may interfere with study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The subject is a non-pregnant female ≥18 years of age, (female sex assigned at birth)
Study Population: Female patients referred for percutaneous coronary intervention (PCI) with coronary IVL and stenting per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2028-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (34):
  - Loma Linda University Health, Loma Linda, California
  - Good Samaritan Hospital, Los Angeles, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - South Denver Cardiology Associates, P.C, Littleton, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory Hospital, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Center for Clinical Research, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New England Heart and Vascular Institute, Manchester, New Hampshire
  - NYU Langone Health, Brooklyn, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Lindner Center for Research and Education at The Christ Hospital CRA: Timothy, Cincinnati, Ohio
  - WellSpan York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MUSC Health University Medical Center, Charleston, South Carolina
  - Centennial Heart, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - DHR Health Heart Institute, McAllen, Texas
  - Baylor Scott & White Research Institute, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - University of Washington Medical Center, Seattle, Washington
- France (4):
  - Centre Hospitalier d'Antibes, Antibes, Antibes
  - Clinique Pasteur, Toulouse, BP 27617
  - AP-HP Hopital Pitie-Salpetriere, Paris, Paris
  - Institut Cardiovasculaire Paris Sud Hôpital Privé Jacques Cartier, Massy
- Germany (3):
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz, Langenbeckstr. 1
  - Krankenhaus der Barmherzigen Bruder Trier, Trier, Nordallee 1
  - Heart and Lung Center Leipzig, Leipzig
- Spain (4):
  - Hospital Clinico De Santiago, Santiago de Compostela, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clínico San Carlos, Madrid
- United Kingdom (4):
  - Golden Jubilee National Hospital, Clydebank
  - Liverpool Heart and Chest Hospital, Liverpool
  - St. George's Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent to Treat: The primary analysis population will be the Intent-to-Treat (ITT) cohort which includes all enrolled subjects.
Period: Overall Study
Arm/Group | Intent to Treat
Started | 399
Completed | 389 (Completed day 30 visit)
Not Completed | 10
Not completed — Death | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Intent-to-Treat (ITT): The primary analysis population will be the Intent-to-Treat (ITT) cohort which includes all enrolled subjects.
Arm/Group | Intent-to-Treat (ITT)
Number analyzed (Participants) | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57
  Not Hispanic or Latino | 299
  Unknown or Not Reported | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Black or African American | 41
  Native Hawaiian or Other Pacific Islander | 0
  White | 319
  Unknown/Not specified | 23
  Other | 5
Subject has Childbearing Potential [Count of Participants; unit: Participants] | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: N=398 because 1 participant did not have a have a height measurement to calculate BMI
  kg/m2
    number analyzed (Participants) | 398
    (all) | 27.9 (5.8)
BMI Categories [Count of Participants; unit: Participants] — Population: N=398 because 1 participant did not have a have a height measurement to calculate BMI
  Participants
    number analyzed (Participants) | 398
    Underweight (below 18.5) | 9
    Healthy weight (18.5 - 24.9) | 126
    Overweight (25 - 29.9) | 140
    Obesity (30 or greater) | 123

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Number of Participants With Target Lesion Failure (TLF) at 30 Days
Description: Target lesion failure (TLF) at 30 days defined as a composite of cardiac death, myocardial infarction (per SCAI definition for peri-procedural MI; per 4th Universal Definition for spontaneous MI beyond discharge) attributable to target vessel (TV-MI), or ischemia-driven target lesion revascularization (ID-TLR).
Time Frame: within 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent-to-Treat (ITT)
Number analyzed (Participants) | 397
Participants | 46

2. Primary Outcome: Primary Effectiveness Endpoint: Procedural Success
Description: Procedural Success defined as stent delivery with a residual in-stent stenosis ≤30% in all target lesions (core laboratory assessed) and without in-hospital TLF (CEC adjudicated).
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat
Number analyzed (Participants) | 390
Participants | 341

3. Secondary Outcome: Angiographic Success (≤30% Residual Stenosis)
Description: Angiographic Success defined as stent delivery with ≤30% residual stenosis and without serious angiographic complications.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Intent to Treat
Number analyzed (Participants) | 390
Number analyzed (Lesions) | 420
Lesions | 407

4. Secondary Outcome: Procedural Success
Description: Procedural Success defined as stent delivery with a residual stenosis <50% in all target lesions (core laboratory assessed) and without in-hospital TLF.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intent to Treat (ITT): The primary analysis population will be the Intent-to-Treat (ITT) cohort which includes all enrolled subjects.
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 390
Participants | 342

5. Secondary Outcome: Angiographic Success (< 50% Residual Stenosis)
Description: Angiographic Success defined as stent delivery with < 50% residual stenosis and without serious angiographic complications.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 390
Number analyzed (Lesions) | 420
Lesions | 408

6. Secondary Outcome: Serious Angiographic Complications
Description: Serious angiographic complications defined as severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 390
Number analyzed (Lesions) | 420
Lesions | 6

7. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: Major Adverse Cardiac Events (MACE) defined as a composite of cardiac death, myocardial infarction (per SCAI definition for periprocedural MI; per 4th Universal Definition for spontaneous MI beyond discharge), and target vessel revascularization. All MACE were adjudicated by an independent CEC.
Time Frame: within 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 397
Participants | 48

8. Secondary Outcome: All Death, Cardiac Death, MI, TV-MI, Procedural and Nonprocedural MI, ID-TVR, ID-TLR, ID-non-TLR, ID-non-TVR, All Revascularizations, and Stent Thrombosis
Description: All death, cardiac death, MI, TV-MI, procedural and nonprocedural MI, ID-TVR, ID-TLR, ID-non-TLR, ID-non-TVR, all revascularizations (ID and non-ID), and stent thrombosis (ARC definite, probable, definite or probable) in-hospital
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 399
Participants
  Death | 4
  Cardiac Death | 3
  MI | 39
  TV-MI | 39
  Procedural MI | 38
  Nonprocedural MI | 1
  ID-TVR | 5
  ID-TLR | 5
  Non-ID-TLR | 0
  Non-ID-TVR | 0
  Revascularizations (ID) | 5
  Revascularizations (non-ID) | 0
  Any Revascularizations | 14
  Stent Thrombosis (ARC definite) | 2
  Stent Thrombosis (ARC probable) | 1
  Stent Thrombosis (ARC definite or probable) | 3

9. Secondary Outcome: All Death, Cardiac Death, MI, TV-MI, Procedural and Nonprocedural MI, ID-TVR, ID-TLR, ID-non-TLR, ID-non-TVR, All Revascularizations, and Stent Thrombosis
Description: All death, cardiac death, MI, TV-MI, procedural and nonprocedural MI, ID-TVR, ID-TLR, ID-non-TLR, ID-non-TVR, all revascularizations (ID and non-ID), and stent thrombosis (ARC definite, probable, definite or probable) through 30 days
Time Frame: within 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 397
Participants
  Death | 8
  Cardiac Death | 4
  MI | 44
  TV-MI | 42
  Procedural MI | 38
  Nonprocedural MI | 8
  ID-TVR | 5
  ID-TLR | 5
  ID-non-TLR | 0
  ID-non-TVR | 0
  Revascularizations (ID) | 5
  Revascularizations (Non-ID) | 0
  Any Revascularizations | 22
  Stent Thrombosis (ARC definite) | 2
  Stent Thrombosis (ARC probable) | 2
  Stent Thrombosis (ARC definite or probable) | 4

10. Secondary Outcome: MI (Myocardial Infarction)
Description: MI rates and all composite endpoints (TLF, MACE) will also be reported using the 4th Universal Definition for peri-procedural and spontaneous MI at all timepoints.
Time Frame: 12-24 hours post procedure or at discharge, whichever is earlier, but at least 4 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 399
Participants
  Peri-procedural MI (<48hrs, SCAI Definition) | 38
  Spontaneous MI (>48hrs, 4th Universal Definition: Type 4a) | 1
  TLF (Target Lesion Failure) | 5

11. Secondary Outcome: MI (Myocardial Infarction)
Description: as for outcome 10
Time Frame: within 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 397
Participants
  Peri-procedural MI (<48hrs, SCAI Definition) | 38
  Spontaneous MI (>48hrs, 4th Universal Definition: Type 4a) | 8
  TLF (Target Lesion Failure) | 46

12. Secondary Outcome: Angina Symptoms Assessed by Seattle Angina Questionnaire (SAQ-7)
Description: Angina symptoms assessed as a change from baseline (at each time period) by Seattle Angina Questionnaire (SAQ-7). Summary score; 0 to 24 represents poor health status; 25 to 49 represents fair; 50 to 74 represents good; 75 to 100 represents excellent.
Time Frame: From baseline to within 30 days of index procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 353
score on a scale | 93.8 [77.5 to 100]

13. Secondary Outcome: Quality of Life Assessed by EQ-5D-5L
Description: Quality of life assessed by EQ-5D-5L as a change from baseline (at each time period). Summary score; ranges from 0-100; 100 represents the best health you can imagine; 0 represents the worst.
Time Frame: From baseline to within 30 days of index procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 352
score on a scale | 7.8 (20.9)

14. Secondary Outcome: Quality of Life Assessed by Generalized Anxiety Disorder Questionnaire (GAD-7)
Description: Quality of life assessed by Generalized Anxiety Disorder Questionnaire (GAD-7) as a change from baseline. Total score calculated by summing points (0-3) for each of the seven questions, yielding a total score from 0-21 (at each time period). Minimal Anxiety (0-4); Mild Anxiety (5-9 ); Moderate Anxiety (10-14 ); Severe Anxiety (≥15).
Time Frame: From baseline to within 30 days of index procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intent to Treat (ITT)
Number analyzed (Participants) | 353
score on a scale | 2.0 [0.0 to 5.0]

ADVERSE EVENTS:
Time Frame: 30 Days
Description: All AE information will be collected from enrollment through the 30 day follow-up visit. Reporting will be carried out in accordance with national regulations. AEs will be followed until the event has resolved (in the case of permanent impairment, the event will be followed until it stabilizes, and the overall clinical outcome has been ascertained). Any AEs that meet IRB/EC reporting requirements must be reported per the institution's policy.
Arm/Group | Intent to Treat (ITT)
All-Cause Mortality (participants affected / at risk) | 8/399
Serious Adverse Events (participants affected / at risk) | 88/399
Other Adverse Events (participants affected / at risk) | 21/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intent to Treat (ITT) (N=399)
Anaemia (Blood and lymphatic system disorders) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 9
Acute myocardial infarction (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 4
Cardiac failure (Cardiac disorders) | 5
Cardiac arrest (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery dissection (Cardiac disorders) | 6
Atrioventricular block complete (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 3
Coronary artery perforation (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Coronary artery thrombosis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Cardiac death (General disorders) | 2
Extravasation (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4
Vascular access site discharge (Injury, poisoning and procedural complications) | 3
Post procedural haematoma (Injury, poisoning and procedural complications) | 2
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
Troponin increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Device malfunction (Product Issues) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
End stage renal disease (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 5
Arterial perforation (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Atherosclerotic plaque rupture (Vascular disorders) | 1
Distributive shock (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intent to Treat (ITT) (N=399)
Angina pectoris (Cardiac disorders) | 11
Vascular access site haematoma (Injury, poisoning and procedural complications) | 10

LIMITATIONS AND CAVEATS:
The study is a post-market observational study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is more than 45 days but less than or equal to 90 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot unilaterally extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT05755711/Prot_SAP_000.pdf